CLINICAL TRIAL: NCT04272788
Title: Association of Breg and Treg With the Clinical Effects of Infliximab in the Treatment of Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2020-01-205
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Infliximab; Treg; Breg
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CD patients: CD patients about to start Infliximab treatment, gives as i.v. injection of 5 mg/kg at baseline, after 2 weeks, 6 weeks, and then every 8th week.CD patients are followed for 14 weeks after the first administration of infliximab. At week 14 of Infliximab treatment, CD patients are classified as remission group (CDAI<150 and endoscopic mucosal healing, R group) and non-remission group (CDAI≥150 and/or mucosal non-healing group, N group).
  Interventions: Drug: Infliximab
- Healthy controls: Healthy controls without Crohn's Disease.

INTERVENTIONS:
Drug: Infliximab — The CD patients at initial active stage without treatment of glucocorticoids, immunosuppressants and biological agents are included in the study when the decision to treat with Infliximab is already made. This study is observational, and all treatment and clinical follow-up are according to national guidelines.
  Groups: CD patients

SUMMARY:
Aims: The main aim of this study is to access the predictive value of Treg and Breg for the clinical effect of Infliximab in the treatment through analyzing the relationship between Breg and Treg and the efficacy of Infliximab.

Design: It is a prospective, observational study. In the treatment group, 32 patients with Crohn's disease (CD) about to start Infliximab-treatment are recruited. They have blood samples drawn at week 0 and 14 of Infliximab treatment. 33 healthy individuals serve as a control group. Controls are only investigated once. All treatment and follow-up are according to national guidelines. The frequencies of Treg and Breg are investigated using flow cytometry. Subjects data are extracted from various registries.

DETAILED DESCRIPTION:
1. Patients with CD at initial active stage are collected from department of gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. The diagnosis of CD is based on clinical, endoscopic, laboratory, radiologic, histo-pathological findings and close follow-up in accordance with the guidelines for the diagnosis and treatment of CD issued by the European Crohn's Disease and Colitis in 2016. Healthy individuals are collected from the Health Examination Center of the Second Affiliated Hospital of Wenzhou Medical University as the healthy controls. The demographic and characteristic information of CD patients and healthy controls are recorded.
2. Infliximab (5mg/kg) is given intravenously at week 0, 2 and 6 to induce CD remission, and then maintained with the same dose of Infliximab every 8 weeks.
3. CD patients are followed for 14 weeks after the first administration of infliximab. At week 14 of Infliximab treatment, according to symptoms, CDAI and endoscopic mucosal healing, CD patients are classified as remission group (CDAI<150 and endoscopic mucosal healing, R group) and non-remission group (CDAI≥150 and/or mucosal non-healing group, N group).
4. C-reactive protein (CRP), leucocyte count (WBC), platelet count (PLT), erythrocyte sedimentation rate (ESR) are detected in CD patients to assess the clinical efficacy at week 0 and 14 of Infliximab treatment respectively.
5. Approximate 5 mL of peripheral fasting venous blood is obtained from every CD patient (at weeks 0 and 14 of Infliximab treatment) and healthy controls. Peripheral blood mononuclear cells (PBMCs) are isolated from the blood samples.
6. Multi-color flow cytometry is applied to examine the frequency of Breg (CD3-CD19+IL-10+ B cell) in B cell: PBMCs are resuspended in RPMI 1640 medium, supplemented with 10% fetal bovine serum and 1% Penicillin/Streptomycin Solution, added in a 96-well flat-bottom culture plate. Then the obtained cells are stimulated with lipopolysaccharide for 48 hours, cultured at 37℃ in 5% CO2 in the incubator, and added Phorbol 12-myristate 13-acetate and ionomycin and Brefeldin A during the final 5 hours. After stimulated and cultured in vitro, PBMCs are stained with FITC-conjugated anti-human CD3 antibodies, APC-conjugated anti-human CD19 antibodies for 30 minutes with blocking light at 4℃. Then stained cells are fixed and permeabilized using a Cytofix/Cytoperm kit and stained with PE-conjugated anti-human IL-10 antibodies for 2 hours at 4℃ that protected form light. Flow staining buffer solution resuspends cells before flow cytometry detection of Breg.
7. Multi-color flow cytometry is applied to examine the frequency of Treg (CD4+CD25+Foxp3+ T cell) in CD4+ T cell: PBMCs are stained with FITC-conjugated anti-human CD4 antibodies, APC-conjugated anti-human CD25 antibodies for 30 minutes with blocking light at 4℃. Stained cells are added fixing buffer and incubated at 4℃ in the dark overnight, then stained with PE-conjugated anti-human FoxP3 antibodies for 2 hours at 4℃ that protected form light. Flow staining buffer solution resuspends cells before flow cytometry detection of Treg.

ELIGIBILITY:
CD patients

Inclusion Criteria:

1. Crohn's Disease at initial active stage with CDAI ≥150.
2. Starting Infliximab treatment

Exclusion Criteria:

1. Significant co-morbidity (e.g. cancer, intestinal tuberculosis, ischemic enteritis, radiation enteritis)
2. Other immunological disease (e.g. diabetes, rheumatoid arthritis systemic lupus erythematosus)
3. Current treatment with glucocorticoids, immunosuppressants and biological agents

Healthy controls

Inclusion Criteria:

1. No current disease
2. No daily drug use

Exclusion Criteria:

1. Significant co-morbidity (e.g. cancer, intestinal tuberculosis, ischemic enteritis, radiation enteritis)
2. Other immunological disease (e.g. diabetes, rheumatoid arthritis systemic lupus erythematosus)
3. Current treatment with glucocorticoids, immunosuppressants and biological agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the gastroenterology department at the Second Affiliated Hospital of Wenzhou Medical University are eligible for entry.
  Healthy controls are recruited at Health Examination Center of the Second Affiliated Hospital of Wenzhou Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Change of the frequency of Treg in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  The frequency of Treg is measured in peripheral blood by flow cytometry.
Change of the frequency of Breg in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  The frequency of Breg is measured in peripheral blood by flow cytometry.
Change of the frequency of Treg in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  The frequency of Treg is measured in peripheral blood by flow cytometry.
Change of the frequency of Breg in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  The frequency of Breg is measured in peripheral blood by flow cytometry.

SECONDARY OUTCOMES:
Change of Crohn's disease activity index (CDAI) in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  CDAI is a measure of Crohn's Disease severity. CDAI < 150 is in remission stage, and ≥ 150 is in active stage. CDAI is negatively correlated with disease activity in CD patients.
Change of C-reactive protein (CRP) in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  CRP is often combined to evaluate the disease activity of CD patients.The normal CRP range is (0-8) mg/L.Increased CRP indicates disease activity.
Change of leucocyte count (WBC) in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  WBC is often combined to evaluate the disease activity of CD patients.The normal WBC range is (4-10)×109/L.Increased WBC indicates disease activity.
Change of platelet count (PLT) in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  PLT is often combined to evaluate the disease activity of CD patients.The normal PLT range is (100-300)×109/L.Increased PLT indicates disease activity.
Change of erythrocyte sedimentation rate (ESR) in R group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  ESR is often combined to evaluate the disease activity of CD patients.The normal ESR range is (0-15)mm/h.Increased ESR indicates disease activity.
Change of Crohn's disease activity index (CDAI) in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  CDAI is a measure of Crohn's Disease severity. CDAI < 150 is in remission stage, and ≥ 150 is in active stage. CDAI is negatively correlated with disease activity in CD patients.
Change of C-reactive protein (CRP) in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  CRP is often combined to evaluate the disease activity of CD patients.The normal CRP range is (0-8) mg/L.Increased CRP indicates disease activity.
Change of leucocyte count (WBC) in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  WBC is often combined to evaluate the disease activity of CD patients.The normal WBC range is (4-10)×109/L.Increased WBC indicates disease activity.
Change of platelet count (PLT) in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  PLT is often combined to evaluate the disease activity of CD patients.The normal PLT range is (100-300)×109/L.Increased PLT indicates disease activity.
Change of erythrocyte sedimentation rate (ESR) in N group | week 0 of Infliximab treatment, week 14 of Infliximab treatment
  ESR is often combined to evaluate the disease activity of CD patients.The normal ESR range is (0-15)mm/h.Increased ESR indicates disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Jiang, PhD, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.